CLINICAL TRIAL: NCT03836339
Title: Appréciation de la Prise en Charge de la Fibrillation Atriale Aux Urgences
Brief Title: Assessment of Atrial Fibrillation in Emergency Department
Acronym: ACFA
Status: Completed | Type: Observational
Sponsor: RESCUe - RESeau Cardiologie Urgence / RESUVal - RESeau des Urgences de la vallée du Rhône (Other)
Collaborators: French Cardiology Society (Other); French Society of Emergency Medicine (Other); Bayer (Industry); Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 2018ACFA10-11
Record Dates: First submitted 2019-01-27; First posted 2019-02-11 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Atrial Fibrillation
Keywords: emergency department; pathway of care; assessment; anticoagulants
MeSH Terms: conditions — Atrial Fibrillation; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Atrial Fibrillation (AF) is the most common disorder of the rhythm disturbance, especially in older adults. The incidence and prevalence of AF increases significantly with age: less than one new case per 1000/year before age 40 to 20/1000 per year after the age of eighty. AF represents 1% of emergency department (ED) visits a third of which are inaugural or recurrent. The causes are varied from cardiac (ischemic cardiac disease, valvular, high blood pressure, heart failure, pericarditis, myocarditis) to extra cardiac etiologies (pulmonary embolism, thyroid disorders, thyrotoxicosis, alcohol, shock, chest trauma, electrolyte disorders, dehydration). While the diagnosis is given quickly by reading the electrocardiogram (ECG), its management both in terms of therapeutic strategy that of choice of care pathway is complex as evidenced by the diversity of possibilities and the difference in practice. Specific recommendations have been published by the French Society of Emergency Medicine in 2015. Our study aims to investigate guidelines implementation in French ED, especially the contribution of diagnostic tests and initiated treatments. Therapeutic strategies are evaluated with a follow up at 3 months, 6 months and 1 year, reporting cardiovascular events and long-term treatment.

DETAILED DESCRIPTION:
This study is non-interventional, recruiting patients presenting to ED with AF. No other epidemiological studies on the subject are available to calculate the required number of subjects and analyze the power of the study. Investigators planned to include 1 575 patients (45 patients in 35 centres) with a minimum targeted 1000 patients to be included in the 30-40 participating centers. The study aims to assess patients characteristics (age, sex, body mass index, type of AF, Congestive Heart failure Hypertension Age Diabetes Stroke - VAscular disease (CHA2DS2- VAsc) Score, Hypertension Abnormal liver/renal function, Stroke history, Bleeding history or predisposition, Labile INR, Elderly, Drug/alcohol usage (HAS-BLED) score), methods of diagnostic (blood tests, ECG, Imaging tests, Cardiac echography), treatment pattern (drugs administered in ED, drug prescribed at hospitalization discharge), patient pathway (orientation after ED admission, discharge, consultation planned), drug-related observance reported by the patient.

Data are collected in a case report form (CRF). Source data verification is performed by sites investigators. A data dictionary containing detailed descriptions of each variable is shared with investigators. Sites monitoring is planned by a clinical research assistant for completing missing data.

Statistical analysis: Data are medians and interquartile ranges (IQRs) for continuous variables, and numbers and percentages for qualitative variables. Stratified analysis of subgroups (age, sex, anticoagulant treatment, examination performed …) will be considered.

ELIGIBILITY:
Inclusion Criteria:

* Atrial fibrillation diagnosis on ECG

Exclusion Criteria:

* Refusal of the patient to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients over 18 years admitted to the emergency department with an AF diagnosis on ECG
Sampling Method: Non-Probability Sample
Enrollment: 1369 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
atrial fibrillation type | At admission
  Number of idiopathic AF, AF secondary to acute heart failure, pulmonary embolism, COPD decompensation, pneumopathy, dysthyroidism, or any other precipitating factor.
Troponin value | At admission
  incidence of positive troponin
Brain Natriuretic Peptide (BNP/proBNP) value | At admission
  incidence of BNP elevation
Renal Clearance | At admission
  Renal clerance(Cl) measuring (by Cockroft formula : Cl(Male) = 1,23 x Weight (kg) x (140 - Age)/Creatinine, Cl(Female) = 1,04 x Weight (kg) x (140 - Age)/Creatinine)
cardiac echography | At admission
  number of cardiac echography performed in ED
antiarythmic drugs | at admission
  list antiarythmic drugs administration (Class IA, IB, IC, II, III or IV of Vaughan Williams classification, digitalis or adenosin)
antiarythmic drugs | at 3 months
  list antiarythmic drugs administration (Class IA, IB, IC, II, III or IV of Vaughan Williams classification, digitalis or adenosin)
antiarythmic drugs | at 6 months
  list antiarythmic drugs administration (Class IA, IB, IC, II, III or IV of Vaughan Williams classification, digitalis or adenosin)
antiarythmic drugs | at 1 year
  list antiarythmic drugs administration (Class IA, IB, IC, II, III or IV of Vaughan Williams classification, digitalis or adenosin)
anticoagulant strategy | at admission
  anticoagulant therapy (vitamin K antagonist or direct oral anticoagulant) administration
anticoagulant strategy | at 3 months, 6 months and 1 year
  anticoagulant therapy (vitamin K antagonist or direct oral anticoagulant) administration
anticoagulant strategy | at 6 months and 1 year
  anticoagulant therapy (vitamin K antagonist or direct oral anticoagulant) administration
anticoagulant strategy | at 1 year
  anticoagulant therapy (vitamin K antagonist or direct oral anticoagulant) administration

SECONDARY OUTCOMES:
mortality | at 24 hours after admission
  number of dead patients
mortality | at 3 months
  number of dead patients
mortality | at 6 months
  number of dead patients
mortality | at 1 year
  number of dead patients
atrial fibrillation incidence | at 3 months
  number of patients with recurrent and persistent
atrial fibrillation incidence | at 6 months
  number of patients with recurrent and persistent
atrial fibrillation incidence | at 1 year
  number of patients with recurrent and persistent
stroke incidence | at admission
  number of new strokes occured
stroke incidence | at 3 months
  number of new strokes occured
stroke incidence | at 6 months
  number of new strokes occured
stroke incidence | at 1 year
  number of new strokes occured
myocardial infarction incidence | at admission
  number of new myocardial infarctions occured
myocardial infarction incidence | at 3 months
  number of new myocardial infarctions occured
myocardial infarction incidence | at 6 months
  number of new myocardial infarctions occured
myocardial infarction incidence | at 1 year
  number of new myocardial infarctions occured
hemorrhagic events | at admission
  type 1, 2 or 3 of the International Society on Thrombosis and Hemostasis classification
hemorrhagic events | at 3 months
  type 1, 2 or 3 of the International Society on Thrombosis and Hemostasis classification
hemorrhagic events | at 6 months
  type 1, 2 or 3 of the International Society on Thrombosis and Hemostasis classification
hemorrhagic events | at 1 year
  type 1, 2 or 3 of the International Society on Thrombosis and Hemostasis classification

CONTACTS AND LOCATIONS:
Overall Officials: Stephane Manzo-Silberman, MD, Principal Investigator — French Cardiology Society
Locations (1):
- Lucien Hussel Hospital, Vienne, France